CLINICAL TRIAL: NCT05254925
Title: Evaluation of Topically Applied Bemotrizinol for Human Phototoxic Potential
Brief Title: Phototoxicity Potential of 6% Bemotrizinol
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: DSM Nutritional Products, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Single | Purpose: Basic Science
Other Study IDs: DSM PT 2020
Record Dates: First submitted 2022-02-11; First posted 2022-02-24 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Phototoxic Response
MeSH Terms: interventions — Sunscreening Agents; bis-ethylhexyloxyphenol methoxyphenyl triazine; Petrolatum

STUDY DESIGN:
Intervention Model Description: The potential of BEMT 6% to produce a phototoxic response will be assessed using a preestablished grading scale for erythema and dermal response following the application of approximately 0.15 g or 0.15 ml of each product (4 investigational treatments) on the skin of human subjects, which will then be exposed to UV radiation. Each study arm will include one of the following investigational treatments: a sunscreen oil with 6% BEMT and 10% ethanol as penetration enhancer (SU E 101413 85) as compared to a Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT (SU E 101413 91); a dispersion of 6% BEMT in petrolatum (SU E 101413 82); and petrolatum vehicle (SU E 101413 83).
Who Masked: Participant
Masking Description: Subjects will be blinded to the name of the investigational products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phototoxicity evaluation of sunscreen oil with 6% BEMT (SU E 101413 85) (Active Comparator): Assessment of the phototoxicity potential of sunscreen oil with 6% BEMT (PARSOL® Shield) and 10% ethanol as penetration enhancer a test material (formulation: SU E 101413 85).
  The phototoxic response of the investigational product: SU E 101413 85 will be assessed following the determination of each subject's Minimal Erythema Dose (MED). Approximately 0.15 g or 0.15 ml of the investigational product will be applied to the skin of human subjects which will then be exposed to UV radiation an a erythema and dermal response scoring system will be used to evaluate the phototoxic response of the irradiated area within the treated test site of each subject.
  Interventions: Drug: Sunscreen oil with 6% Bemotrizinol
- Phototoxicity evaluation of sunscreen oil vehicle (SU E 101413 91) (Other): Vehicle Control: Assessment of the phototoxicity potential of sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT (formulation: SU E 101413 91).
  The phototoxic response of the investigational product: SU E 101413 91 will be assessed following the determination of each subject's Minimal Erythema Dose (MED). Approximately 0.15 g or 0.15 ml of the investigational product will be applied to the skin of human subjects which will then be exposed to UV radiation an a erythema and dermal response scoring system will be used to evaluate the phototoxic response of the irradiated area within the treated test site of each subject.
  Interventions: Other: Sunscreen oil vehicle
- Phototoxicity evaluation of dispersion of 6% BEMT in petrolatum (SU E 101413 82) (Active Comparator): Assessment of the phototoxicity potential of a dispersion of 6% BEMT (PARSOL® Shield) in petrolatum (formulation: SU E 101413 82).
  The phototoxic response of the investigational product: SU E 101413 82 will be assessed following the determination of each subject's Minimal Erythema Dose (MED). Approximately 0.15 g or 0.15 ml of the investigational product will be applied to the skin of human subjects which will then be exposed to UV radiation an a erythema and dermal response scoring system will be used to evaluate the phototoxic response of the irradiated area within the treated test site of each subject.
  Interventions: Drug: Dispersion of 6% BEMT in petrolatum
- Phototoxicity evaluation of petrolatum vehicle (SU-E-101413-83) (Other): Vehicle Control: Assessment of the phototoxicity potential of petrolatum vehicle (SU-E-101413-83).
  The phototoxic response of the investigational product: SU E 101413 83 will be assessed following the determination of each subject's Minimal Erythema Dose (MED). Approximately 0.15 g or 0.15 ml of the investigational product will be applied to the skin of human subjects which will then be exposed to UV radiation an a erythema and dermal response scoring system will be used to evaluate the phototoxic response of the irradiated area within the treated test site of each subject.
  Interventions: Other: Petrolatum vehicle

INTERVENTIONS:
Drug: Sunscreen oil with 6% Bemotrizinol — Sunscreen oil with 6% BEMT (PARSOL® Shield) and 10% ethanol as penetration enhancer
  Other Names: PARSOL® SHIELD; SU E 101413 85
  Arms: Phototoxicity evaluation of sunscreen oil with 6% BEMT (SU E 101413 85)
Other: Sunscreen oil vehicle — Sunscreen oil vehicle with 10% ethanol as penetration enhancer without BEMT (BEMT replaced by Isopropylmyristate)
  Other Names: SU E 101413 91
  Arms: Phototoxicity evaluation of sunscreen oil vehicle (SU E 101413 91)
Drug: Dispersion of 6% BEMT in petrolatum — Dispersion of 6% BEMT (PARSOL® Shield) in petrolatum
  Other Names: PARSOL® SHIELD; SU-E-101413-82
  Arms: Phototoxicity evaluation of dispersion of 6% BEMT in petrolatum (SU E 101413 82)
Other: Petrolatum vehicle — Petrolatum vehicle
  Other Names: SU-E-101413-83
  Arms: Phototoxicity evaluation of petrolatum vehicle (SU-E-101413-83)

SUMMARY:
Phototoxicity Potential of Bemotrizinol (6%)

DETAILED DESCRIPTION:
This clinical trial will assess the phototoxic potential of a test material, compared to a vehicle control and a negative control. The results obtained will determine if 6% bemotrizinol (BEMT) either in a basic sunscreen oil formulation SU E 101413 85 or as dispersion in petrolatum (SU-E-101413-82) elicit a phototoxic response based on a comparison of the reactions obtained (either Phototoxic or non-Phototoxic) on the treated/irradiated, treated/non-irradiated and non- treated control sites. Two vehicle controls, i.e. sunscreen oil vehicle (SU E 101413 91) and petrolatum (SU E 101413 83), and a negative control will also be used as comparators in this clinical trial.

Duplicate test sites on the back (each approximately 4 cm2) will be identified via use of body map demonstrating application sites. Test material will be applied to designated patches and affixed to both sides of the back. In addition, 2 sets of patches without test material will be applied on 2 sides of the back. One side will be designated for irradiation, and the other is used as a treated/non-irradiated, and non-treated/non- irradiated control.

Approximately 24 hours after application, the patches will be removed and the skin will be gently wiped. The Minimal Erythema Dose (MED) will be determined from the five UV-treated sub-sites and all of the test sites will be evaluated according to the erythema grading scale. For evaluation of phototoxicity, the sites are irradiated with 0.5 of the subject's MED (full spectrum wavelengths UVB 290-320 nm and UVA 320-400 nm) followed by 5 J/cm2 UVA (320-400nm) using a Schott WG-345 and UG11/1 mm filter to block UVB wavelength 290-320 nanometers. The sites designated for irradiation will be then irradiated with solar simulated light by 0.5 times an individual's MED followed by 5 J/cm2 UVA.

Statistical analysis will not be performed for this study. Investigational product safety will be determined through interpretation of the dermal evaluation scores. Treated and control sites will be examined at 24 and 48 hours post-irradiation and graded according to a scoring scale.

If a grade ≥2+ erythema is observed after patch removal on the site designated for irradiation, the site will not be irradiated, regardless of the dermal response of the non-irradiated site and the subjects will be discontinued by the Principal Investigator from the study. The dermal response will be followed up until resolution or until the end of the study.

Dermal scores will be reported for each site. Clinically significant reactions other than phototoxic reactions will be recorded and interpreted accordingly and the safety of the investigational product will be monitored by evaluating adverse event reporting. An adverse event is any untoward medical occurrence, whether or not it is considered clinical trial related, including death, experienced by a subject. An event may consist of a disease, an exacerbation of a pre-existing illness or condition, an occurrence of an intermittent illness or condition, a set of related symptoms or signs, or a single symptom or sign. Any subject that presents with a dermal reaction of 3+ or greater will be considered as an adverse event and documented accordingly.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female between 18 and 75 years of age;
2. Subject has a Fitzpatrick Skin Types I - III, based on the first 30 to 45 minutes of sun exposure after a winter season of no sun exposure according to the following criteria; I Always burns easily; never tans (sensitive) II Always burns easily; tans minimally (sensitive) III Burns moderately; tans gradually (normal)
3. Subject agrees to avoid excessive sun exposure of the test sites and to refrain from visits to tanning salons during the course of this study;
4. Subject does not exhibit any skin diseases or abnormalities which might be confused with a skin reaction from the test material;
5. Subject agrees not to introduce any new cosmetic or toiletry products during the study;
6. Subject agrees to refrain from getting patches wet and from scrubbing or washing the test area with soap or applying powders, lotions or personal care products to the area during the course of the study;
7. Subject is dependable and able to follow directions as outlined in the protocol and anticipates being available for all study visits;
8. Subject is willing to participate in all study evaluations;
9. Subject is in generally good health and has a current Panelist Profile Form on file at CRL;
10. Subject has completed a HIPAA Authorization Form in conformance with 45 CFR Parts 160 and 164;
11. Subject understands and is willing to sign an Informed Consent Form in conformance with 21 CFR Part 50: "Protection of Human Subjects."

Exclusion Criteria:

1. Female subject is pregnant, nursing, planning a pregnancy, or not using adequate birth control;
2. Subjects with a prior history of phototoxic or photoallergic reactions or those taking medication which might produce an abnormal response to sunlight;
3. Subject has received treatment with sympathomimetics, antihistamines, vasoconstrictors, non-steroidal anti-inflammatory agents, and/or systemic or topical corticosteroids within one week prior to initiation of the study;
4. Subject has a history of acute or chronic dermatologic, medical, and/or physical conditions which would preclude application of the test material and/or could influence the outcome of the study;
5. Subject is under treatment for a skin and/or systemic bacterial infection;
6. Subject reports a history of allergies to tape adhesives;
7. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
8. Subject has known allergies to sunscreen, skin treatment products or cosmetics, toiletries, and/or topical drugs;
9. Subject has a known communicable disease (e.g., HIV, sexually transmitted diseases, Hepatitis B, Hepatitis C, etc.);
10. Subject has insulin-dependent diabetes;
11. Subject has a history of cancer;
12. Subject is currently taking certain medications which, in the opinion of the Principal Investigator, may interfere with the study;
13. Subject exhibits sunburn, suntan, uneven skin tone, blemishes, moles or excess hair in the test site area.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-04-03 (Actual)

PRIMARY OUTCOMES:
Determination of the Photoxicity potential of 6% Bemotrizinol 24 hours post-irradiation | Phototoxic response will be checked 24 hours post-irradiation
  Phototoxic response based on a comparison of the reactions obtained on treated/irradiated, treated/non-irradiated and non-treated control sites
  Investigational product safety will be determined through interpretation of the dermal evaluation scores. Dermal scores will be reported as either Phototoxic or Non-Phototoxic responses and the following dermal scoring system will be used to evaluate the irradiated area within the treated test site:
  Grading scale for Erythema:
  "0" = No visible skin reaction; "+" = Barely perceptible erythema; "1+" = Mild erythema; "2+" = Well defined erythema; "3+" = Severe erythema
  Grading Scale for dermal response:
  e = Edema P = Peeling S = Spreading of reaction beyond irradiated site. Sc = Scabbing d = Dryness/scaling D = Oozing, crusting, and/or superficial erosions I = Itching Pa = Papules V = Vesicle W = Weeping Hr = Hyperpigmentation Ho = Hypopigmentation M = Missed Visit
Determination of the Photoxicity potential of 6% Bemotrizinol 48 hours post-irradiation | Phototoxic response will be checked 48 hours post-irradiation
  Phototoxic response based on a comparison of the reactions obtained on treated/irradiated, treated/non-irradiated and non-treated control sites
  Investigational product safety will be determined through interpretation of the dermal evaluation scores. Dermal scores will be reported as either Phototoxic or Non-Phototoxic responses and the following dermal scoring system will be used to evaluate the irradiated area within the treated test site:
  Grading scale for Erythema:
  "0" = No visible skin reaction; "+" = Barely perceptible erythema; "1+" = Mild erythema; "2+" = Well defined erythema; "3+" = Severe erythema
  Grading Scale for dermal response:
  e = Edema P = Peeling S = Spreading of reaction beyond irradiated site. Sc = Scabbing d = Dryness/scaling D = Oozing, crusting, and/or superficial erosions I = Itching Pa = Papules V = Vesicle W = Weeping Hr = Hyperpigmentation Ho = Hypopigmentation M = Missed Visit

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Schutz, PhD, Study Director — DSM Nutritional Products, Inc.; Gladys Osis, MT, Principal Investigator — Eurofins CRL Inc.
Locations (1):
- Eurofins | CRL, Inc., Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No